CLINICAL TRIAL: NCT06049602
Title: Efficacy of TDF and Entekavir Prophylaxis at Hepatitis B Reactivation: Multi Center Retrospective Study
Brief Title: TDF and Entekavir - Hepatitis B Reactivation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Viral Hepatitis Society (Other)
Responsible Party: Sponsor
Other Study IDs: IMMUNHEP
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hepatitis B Reactivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional retrospective multi-center study for the patients received Entekavir or TDF for Hepatitis B prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patients used entekavir or TDF for Hepatitis B prophylaxis

Exclusion Criteria:

* Patients lower then 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who used entekavir or TDF for Hepatitis B prophylaxis
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Reactivation Rate | 12 months
  Percentage of patients reactivated during the Entekavir or TDF

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Kurkcu, Study Director — Sentez CRO
Locations (1):
- Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No